CLINICAL TRIAL: NCT04117113
Title: Prospective Epidemiological Study to Estimate the O-serotype Distribution of Extraintestinal Pathogenic Escherichia Coli (ExPEC) Isolated From Hospitalized Patients Aged 60 Years or Older With Invasive ExPEC Disease (IED) and to Evaluate the Clinical Case Definition and Risk Factors.
Brief Title: Study to Collect Information About Invasive Disease Caused by Extraintestinal Pathogenic Escherichia Coli-2 (EXPECT-2)
Acronym: EXPECT-2
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Janssen Research & Development, LLC (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Principal Investigator, MJM Bonten, Professor of Molecular Epidemiology of Infectious Diseases, UMC Utrecht
Other Study IDs: VAC52416BAC0006
Record Dates: First submitted 2019-05-22; First posted 2019-10-07 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: E. Coli Infection
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — E. coli isolates from blood, urine, or any other normally sterile body site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly, 60+ hospitalized with Invasive ExPEC Disease: Patients 60 years or older hospitalized with Invasive Extraintestinal Pathogenic Escherichia coli Disease.

SUMMARY:
The purpose of this study is to collect information from study participants who are hospitalized with an invasive disease caused by Extraintestinal pathogenic E. coli (ExPEC). This information will be used to support the development of a new vaccine to prevent Extraintestinal pathogenic Escherichia coli (ExPEC). E. coli bacteria are a leading cause of serious infections. Especially adults older than 60 years have a higher risk of developing such infections. To date, there is no vaccine available to prevent E. coli infections. To support the development of a vaccine, more information about E. coli infections is first needed. This information will be collected in the current study, such as:

* Medical information such as medical history, diagnosis, duration of hospitalization
* Treatment and outcome of the Extraintestinal pathogenic Escherichia coli (ExPEC)
* Laboratory information

DETAILED DESCRIPTION:
Janssen Research & Development is developing ExPEC10V, a 10-valent conjugate vaccine comprising the 10 most predominant O-polysaccharides of ExPEC.

Invasive ExPEC Disease (IED) is defined as an acute illness consistent with bacterial infection that is microbiologically confirmed either by the isolation and identification of E. coli from blood or other normally sterile body sites, or by the isolation and identification of E. coli from urine in a patient with signs and symptoms of invasive disease (presence of systemic inflammatory response syndrome [SIRS], sepsis or septic shock) and no other identifiable source of infection.

ExPEC is the most common cause of infection in humans resulting from gram-negative bacteria. ExPEC comprises a pathogenic group of E. coli strains, possessing the ability to colonize and infect normally sterile body sites and to cause Invasive ExPEC Disease (IED).

ExPEC causes the vast majority of urinary tract infections (UTIs), is the second most frequent cause of neonatal bacteremia and meningitis, and is a leading cause of adult IED, in particular bacteremia and sepsis.

Although IED affects all age categories, adults aged 60 years or older have an increased risk of developing IED, including bacteremia and sepsis. The incidence of community-acquired ExPEC bacteremia increases with age, occurring at a rate of 150/100,000 person-years in the United States (US) adults aged 65 years and older, and 452/100,000 person-years in adults aged 85 years and older. Similar trends have been observed in Europe. In the US, it is estimated that up to 40,000 patients die annually due to IED, in particular from E. coli sepsis. Overall case-fatality rates for ExPEC bacteremia range from 13% to 19% but may be much higher (up to 60%) in the elderly with healthcare-associated infections.

The increase in multidrug resistance (ie, resistance to two or more antibiotic classes) among ExPEC strains, such as E. coli sequence type 131:O25B, represents a major challenge for prevention and management of ExPEC infections. Global morbidity, hospitalization and mortality rates due to ExPEC infections are substantial and increasing due to aging populations and increasing prevalence of antibiotic resistant ExPEC strains, and associated with increasing healthcare costs in both Europe and the US.

This hospital-based prospective epidemiological study will assess the O-serotype and O-genotype distribution in E. coli isolates causing IED overall and by subgroup based on risk factors. Detailed demographic and clinical data, including information on hospital routes, from patients with IED will be collected in this study to further characterize the clinical setting in this patient population. This study will also provide data to compare the clinical criteria of IED used by the study site with the proposed Phase 3 clinical case definition for IED in adults aged 60 years or older for future clinical studies in this patient population. No study drug will be administered in this non interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or older and hospitalized for IED at the start of the study.
* Culture confirmation of E. coli (1) in normally sterile body sites including blood, and/or (2) in urine in the presence of clinical criteria of an invasive infection (raise in SOFA score >1, sepsis, or septic shock consequent to the infection).
* For those countries and/or study sites where no waiver for informed consent/assent has been obtained prior to data collection, eligible patients must sign a participation agreement/ICF/IAF allowing data collection and source data verification in accordance with local requirements and/or sponsor policy. For deceased patients, a participation agreement/ICF/IAF must be signed by the patient's next of kin.

Exclusion Criteria:

• There are no exclusion criteria for this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized and having culture-confirmed IED.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Distribution of E. coli O-serotypes causing IED in adults aged 60 years or older, as percentage of the total study population. | 12 months
Distribution of E. coli O-genotypes causing IED in adults aged 60 years or older, as percentage of the total study population. | 12 months
Distribution of IED in adults aged 60 years or older over the following clinical case definitions: "Pyelonephritis", "Urosepsis", "Meningitis", "Arthritis", "Sepsis of unknown origin" and "Others", as a percentage of the total study population. | 12 months

SECONDARY OUTCOMES:
Proportion of non-bacteremic and bacteremic IED of the total number of IED cases. | 12 months
Listing of IED patients with specific risk factors for IED as a proportion of all IED patients. | 12 months
  Specific risk factors for IED are medical conditions (e.g. kidney disease, history of urinary tract infection in prior 12 months), sociodemographic characteristics (e.g. age, gender) and medication use (e.g. immunosuppressive medication)
Type of infection (community acquired, hospital-acquired or healthcare-associated) . | 12 months
Source of infection (presence of an infectious focus within 30 days prior to IED). | 12 months
Susceptibility of the cultured E. coli strains to antibiotics as determined by EUCAST standards (version9.0) to β-lactam antibiotics. | 12 months
O-antigen expression profiles | 12 months
Mortality associated with IED | 12 months
Department where patient is presented/admitted to the hospital (emergency ward, general ward, intensive care unit) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Miquel B Ekkelenkamp, MD, Principal Investigator — UMC Utrecht
Locations (8):
- Duke Clinical Research Institute, Durham, North Carolina, United States
- Duke Clinical Research Institute, Greater Sudbury, Canada
- CHU Limoges - CIC, Limoges, France
- UKK Uniclinic Cologne, Cologne, Germany
- University of Verona, Verona, Italy
- Janssen Pharmaceutical K.K., Tokyo, Chiyoda-ku, Japan
- Andalusian Public Foundation for Health Research Management in Seville (FISEVI), Seville, Spain
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No